CLINICAL TRIAL: NCT00193310
Title: Preoperative (Neoadjuvant) or Postoperative (Adjuvant) Therapy of Patients With Stages IB, II, IIIA Non-Small Cell Lung Cancer
Brief Title: Preoperative or Postoperative Therapy of Patients With Stages IB, II, IIIA Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 53
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Paclitaxel; Carboplatin

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
In this phase II study, we plan to evaluate several novel components of therapy. In patients with potentially resectable stages IIB (T3N0) and IIIA we will compare weekly paclitaxel and carboplatin with concomitant radiation therapy versus weekly paclitaxel and every 4 week carboplatin in the preoperative (neoadjuvant) setting. For patients with potentially resectable stage IB, IIA and IIB (T2N1) tumors, weekly paclitaxel and every 4 week carboplatin will be given pre-operatively (neoadjuvant). The feasibility of resection will be evaluated in the neoadjuvant group of patients. The continued study of concurrent radiation therapy with weekly paclitaxel and carboplatin will be evaluated in those patients with stage IIB (T3N0) and IIIA disease who initially had resection (adjuvant setting). Lastly, weekly paclitaxel and carboplatin every 4 weeks will be evaluated as an adjuvant program in patients who had completely resected stage IB, IIA and IIB (T2N1).

DETAILED DESCRIPTION:
Upon determination of eligibility, neo-adjuvant patients will be randomly assigned to one of two treatment arms:

* ARM A Paclitaxel + Carboplatin + Radiation Therapy + Surgery
* ARM B Paclitaxel + Carboplatin + Surgery

After surgery neo-adjuvant patients with a complete resection will either receive Paclitaxel + Carboplatin or no therapy, depending on their stage of disease at time of enrollment. Patients with incomplete resection Paclitaxel + Carboplatin + Radiation Therapy. Adjuvant patients who enter the study after complete resection will receive Paclitaxel + Carboplatin with or without Radiation Therapy based on initial stage of disease.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Non-small cell lung cancer
* Neoadjuvant candidates must have potentially resectable disease
* Adjuvant candidates must have had complete resection
* Clinical stage IB, II, or IIIA non-small cell lung cancer
* ECOG performance status 0 or 1
* Adequate bone marrow, liver and kidney function
* No previous chemotherapy or radiation therapy for non-small cell lung cancer.
* Give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Stage IIIA with N2 nodes > 6 cm
* Stage IIIB or IV disease
* Age <18 years
* ECOG performance status 2 or higher
* Considered inoperable based on general medical condition
* History of prior malignancy within five years
* Women who are pregnant or lactating

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2000-11; Primary Completion 2003-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall response rates

SECONDARY OUTCOMES:
Resectability rates
Survival
Time to progression
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Greco, MD, Principal Investigator — SCRI Development Innovations, LLC